CLINICAL TRIAL: NCT02406937
Title: Efficacy of New Stage 1 Formula on the Improvement of Gut Comfort and Gut Health
Brief Title: New Stage 1 Formula on Gut Comfort and Gut Health
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heilongjiang Feihe Dairy Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14-SC-9-FH-001
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Lactation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Feihe New Formula (Experimental): Oral intake of Feihe new formula with hydrolyzed protein supplied by Arla Foods Ingredients.
  Interventions: Dietary Supplement: Oral intake of Feihe New Formula
- Feihe Stage 1 Formula (Active Comparator): Oral intake of Feihe stage 1 formula
  Interventions: Dietary Supplement: Oral intake of Feihe Stage 1 Formula
- Breast Feeding (Placebo Comparator): Oral intake of breast milk
  Interventions: Dietary Supplement: Breast Feeding

INTERVENTIONS:
Dietary Supplement: Oral intake of Feihe New Formula — Oral intake of Feihe New Formula
  Arms: Feihe New Formula
Dietary Supplement: Oral intake of Feihe Stage 1 Formula — Oral intake of Feihe Stage 1 Formula
  Arms: Feihe Stage 1 Formula
Dietary Supplement: Breast Feeding — Oral intake of breast milk
  Arms: Breast Feeding

SUMMARY:
180 qualified subjects aged from 7 days to 90 days will be enrolled with the 144 completed in study (allowing for a 20% drop-out rate). Subjects will be randomly assigned into 3 groups, including breast feeding, commercial and new formula group. Study intervention is 12 weeks.

DETAILED DESCRIPTION:
Primary objective:

1. Improvement on gut health and infant comfort

Secondary objective：

1. Efficacy on easy digestion;
2. Changes on SCFA in feces(Baseline and Endpoint)
3. Improvement on gut microbiome strains(Baseline and Day 21); (bifidobacterium/lactobacillus/clostridium perfringens recommended)
4. Changes on sIgA in feces(Baseline and Endpoint)
5. Improvement on tolerance(comfort) via infant fussy/bloating/abdominal pain/milk regurgitation/sleeping time;
6. Incidence of eczema and duration;
7. Infants growth

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 7-90 days;
* Fed by breast milk before enrollment;
* Parent or legal guardian fully understand the purpose and requirement, including the potential risks and side effects of the study;
* Willing to participate in the study and comply all the procedures;
* Concent form signed by parents.

Exclusion Criteria:

* Twins, multiple birth, low birth weight children, over birth weight children or early birth children with gestational age less than 37 weeks;
* Think about the need to exclude C-section delivered infants? It's often the majority of births in Chinese tier-1 cities, so it will probably make the study recruitment slower, and postpone the study. The microflora of C-section infants in known to be different compared to normally born infants. At least, the mode of delivery should be noted and calculated into the primary and secondary outcome measurements as a potential confounding factor
* During pregnancy, the mothers had pregnancy complications or other disease that may affect the results;
* Having serious diseases that may affect study interventions, such as neonatal sepsis, pneumonia (associated with respiratory failure), heart failure and other disease;
* Having neonatal diarrhea or acute respiratory infections within 48hours before enrollment;
* Having potential metabolic diseases, chronic diseases, congenital malformations, central nervous system disorders, neuromuscular disorders or diseases affecting bone metabolism that may affect growth or the study results;
* Having taken any food containing prebiotics or probiotics tithing 15 days of enrollment;
* Having gluten allergy (celiac disease);
* Body weight-to-height Z-value<-3 according to the standard of WHO;
* Receiving hormone therapy and intravenous nutrition;
* Lactose intolerance or allergic to ingredients of study product;
* Have participated in other clinical studies within 3 months prior to the date of screening;
* Unable to comply the study schedule.

Ages: 7 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiancun Pan, Study Director — Heilongjiang Feihe Dairy Co. Ltd.
Locations (1):
- Sprim (Shanghai) Consulting Co., Ltd., Shanghai, Shanghai Municipality, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Feihe New Formula: Oral intake of Feihe new formula with hydrolyzed protein supplied by Arla Foods Ingredients.
  Oral intake: Oral intake
- Feihe Formula: Oral intake of Feihe stage 1 formula
  Oral intake: Oral intake
- Breast Feeding: Oral intake of breast milk
  Oral intake: Oral intake
Period: Overall Study
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Started | 60 | 60 | 60
Completed | 59 | 59 | 58
Not Completed | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding | Total
Number analyzed (Participants) | 59 | 59 | 58 | 176
Age, Continuous [Mean (Standard Deviation); unit: Days] | 55.5 (18.3) | 58.4 (17.0) | 59.8 (20.5) | 57.9 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 24 | 83
  Male | 29 | 30 | 34 | 93
Region of Enrollment [Number; unit: participants]
  China | 59 | 59 | 58 | 176

OUTCOME MEASURES:

1. Primary Outcome: Stool Frequency
Description: Average daily stool frequency during the measurement week
Time Frame: Baseline, Week 4, Week 8, Week 12
Measure: Mean (Standard Deviation); unit: Times per day
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
Times per day
  Baseline | 2.2 (1.0) | 2.2 (0.9) | 2.3 (1.0)
  Week 4 | 1.6 (0.5) | 1.8 (0.6) | 2.1 (0.7)
  Week 8 | 1.2 (0.3) | 1.6 (0.5) | 1.5 (0.5)
  Week 12 | 1.0 (0.3) | 1.5 (0.4) | 1.6 (0.4)

2. Secondary Outcome: Number of Participants With Gastrointestinal Symptoms
Description: Number of participants with symptom of bloating and abdominal pain
Time Frame: Weekly (Baseline to Day 84)
Measure: Number; unit: participants
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
participants | 0 | 0 | 0

3. Secondary Outcome: Stool Consistency
Description: Average Bristol Score during the measurement week. The seven types of stool are:
  1. = Separate hard lumps, like nuts (difficult to pass)
  2. = Sausage-shaped but lumpy
  3. = Like a sausage but with cracks in its surface
  4. = Like a sausage or snake, smooth and soft
  5. = Soft blobs with clear-cut edges (passed easily)
  6. = Fluffy pieces with ragged edges; a mushy stool
  7. = Watery, no solid pieces, entirely liquid Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools (especially the latter), as they are easy to defecate while not containing excess liquid, and 5, 6 and 7 tending towards diarrhoea.
Time Frame: Baseline, Week 4, Week 8, Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
units on a scale
  Baseline | 3.61 (0.63) | 3.74 (0.55) | 3.76 (0.90)
  Week 4 | 3.19 (0.63) | 3.59 (0.50) | 3.73 (0.66)
  Week 8 | 3.09 (0.44) | 3.38 (0.38) | 3.50 (0.51)
  Week 12 | 3.05 (0.79) | 3.35 (0.46) | 3.57 (0.62)

4. Secondary Outcome: Crying Time
Description: Questionnaire recorded by parents. Average crying time per day during the measurement week.
Time Frame: Baseline, Week 4, Week 8, Week 12
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
minutes/day
  Baseline | 2.98 (2.88) | 2.90 (1.65) | 2.92 (2.65)
  Week 4 | 3.43 (1.37) | 2.69 (0.97) | 2.62 (2.26)
  Week 8 | 2.72 (0.77) | 2.40 (0.69) | 2.34 (1.02)
  Week 12 | 2.83 (0.79) | 2.06 (0.56) | 2.01 (0.48)

5. Secondary Outcome: Fecal Concentration of Short Chain Fatty Acid
Description: fecal concentration of acetate, propionate and butyrate acid
Time Frame: Baseline, Day 21
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
mg/g
  Baseline acetate acid | 4.66 (1.31) | 4.75 (1.57) | 4.72 (1.73)
  Baseline propionate acid | 1.28 (0.51) | 1.27 (0.61) | 1.33 (0.60)
  Baseline butyrate acid | 0.83 (0.51) | 0.85 (0.46) | 0.81 (0.57)
  Day 21 acetate acid | 4.14 (1.10) | 4.77 (1.50) | 4.88 (1.93)
  Day 21 propionate acid | 1.32 (0.52) | 1.35 (0.51) | 1.42 (0.68)
  Day 21 butyrate acid | 0.84 (0.49) | 0.87 (0.47) | 0.86 (0.61)

6. Secondary Outcome: Body Length
Description: Body length
Time Frame: Baseline, Day 28, Day 56, Day 84
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
cm
  Baseline | 56.9 (2.3) | 57.7 (2.4) | 57.8 (2.8)
  Day 28 | 60.3 (2.2) | 60.8 (2.2) | 61.1 (2.7)
  Day 56 | 62.6 (2.0) | 63.2 (2.3) | 63.5 (2.3)
  Day 84 | 64.6 (2.2) | 64.8 (2.4) | 65.4 (2.3)

7. Secondary Outcome: Number of Participants With Eczema
Time Frame: Throughout the study period (84 days)
Measure: Number; unit: participants
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
participants | 15 | 9 | 8

8. Secondary Outcome: Fecal Laboratory Detection for sIgA
Time Frame: Baseline, Day 84
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
ug/ml
  Baseline | 53.8 (19.5) | 53.0 (20.7) | 55.5 (20.3)
  Day 84 | 55.3 (12.9) | 62.7 (11.8) | 65.9 (10.8)

9. Secondary Outcome: Fecal Bacterium Concentration
Description: bifidobacterium, lactobacillus, clostridium perfringens
Time Frame: Baseline, Day 21
Measure: Mean (Standard Deviation); unit: log (colony forming units)
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
log (colony forming units)
  Baseline bifidobacterium | 7.56 (0.76) | 7.55 (0.71) | 7.58 (0.75)
  Baseline lactobacillus | 6.61 (0.86) | 6.58 (0.83) | 6.63 (0.78)
  Baseline clostridium perfringens | 4.69 (1.28) | 4.73 (1.20) | 4.64 (1.20)
  Day 21 bifidobacterium | 7.51 (0.55) | 7.67 (0.53) | 7.71 (0.65)
  Day 21 lactobacillus | 6.65 (0.95) | 6.78 (0.98) | 6.80 (0.82)
  Day 21 clostridium perfringens | 4.73 (1.26) | 4.57 (1.41) | 4.51 (1.51)

10. Secondary Outcome: Eczema Duration
Time Frame: Throughout the study period (84 days)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
Days | 62.1 (15.0) | 45.2 (21.1) | 38.6 (17.6)

11. Secondary Outcome: Body Weight
Time Frame: Baseline, Day 28, Day 56, Day 84
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
g
  Baseline | 5191.5 (715.2) | 5291.5 (738.9) | 5462.1 (1040.0)
  Day 28 | 6142.4 (678.3) | 6251.7 (747.5) | 6370.7 (912.1)
  Day 56 | 6922.9 (701.5) | 6975.4 (712.9) | 7102.6 (842.5)
  Day 84 | 7430.5 (650.0) | 7484.1 (699.1) | 7575.0 (775.6)

12. Secondary Outcome: Head Circumference
Time Frame: Baseline, Day 28, Day 56, Day 84
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
cm
  Baseline | 38.5 (1.2) | 38.7 (1.2) | 39.0 (1.3)
  Day 28 | 39.9 (1.1) | 40.1 (1.1) | 40.4 (1.2)
  Day 56 | 41.1 (1.0) | 41.4 (1.1) | 41.5 (1.2)
  Day 84 | 42.1 (1.0) | 42.4 (1.0) | 42.4 (1.0)

13. Secondary Outcome: Chest Circumference
Time Frame: Baseline, Day 28, Day 56, Day 84
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
cm
  Baseline | 36.9 (1.2) | 37.2 (1.1) | 37.3 (1.3)
  Day 28 | 38.2 (1.1) | 38.6 (1.2) | 38.7 (1.3)
  Day 56 | 39.4 (1.0) | 39.6 (1.1) | 39.8 (1.2)
  Day 84 | 40.5 (1.0) | 40.6 (1.0) | 40.9 (1.0)

14. Secondary Outcome: Milk Regurgitation Frequency
Description: Questionnaire recorded by parents. Average daily frequency of milk regurgitation during the measurement week.
Time Frame: Baseline, Week 4, Week 8, Week 12
Measure: Mean (Standard Deviation); unit: Times/day
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
Times/day
  Baseline | 2.68 (1.60) | 2.47 (1.42) | 2.43 (1.74)
  Week 4 | 2.70 (1.27) | 2.02 (0.89) | 1.89 (1.25)
  Week 8 | 1.75 (1.21) | 1.25 (0.61) | 1.17 (0.84)
  Week 12 | 1.05 (0.79) | 0.71 (0.40) | 0.64 (0.60)

15. Secondary Outcome: Milk Feeding Quantity
Description: Questionnaire recorded by parents. Average quantity of milk feeding per day during the measurement week.
Time Frame: Baseline, Week 4, Week 8, Week 12
Measure: Mean (Standard Deviation); unit: ml/day
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
ml/day
  Baseline | 732.1 (169.3) | 742.2 (97.6) | 750.7 (119.4)
  Week 4 | 928.6 (104.6) | 936.3 (88.3) | 946.0 (98.4)
  Week 8 | 1063.3 (107.1) | 1062.0 (98.1) | 1070.2 (83.3)
  Week 12 | 1179.0 (101.5) | 1181.8 (95.0) | 1182.9 (69.6)

16. Secondary Outcome: Sleeping Time
Description: Questionnaire recorded by parents. Average sleeping time per day during the measurement week.
Time Frame: Baseline, Week 4, Week 8, Week 12
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
hours/day
  Baseline | 18.0 (0.8) | 17.8 (0.6) | 17.9 (1.3)
  Week 4 | 17.6 (0.8) | 17.4 (0.5) | 17.6 (0.9)
  Week 8 | 16.9 (0.5) | 16.8 (0.5) | 16.9 (0.4)
  Week 12 | 16.4 (0.6) | 16.4 (0.5) | 16.5 (0.6)

17. Secondary Outcome: Body Mass Index (BMI)
Description: BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m^2 (kilogram per square meter).
Time Frame: Baseline, Week 4, Week 8, Week 12
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Feihe New Formula | Feihe Stage 1 Formula | Breast Feeding
Number analyzed (Participants) | 59 | 59 | 58
kg/m^2
  Baseline | 15.9 (1.3) | 15.8 (1.4) | 16.2 (1.7)
  Week 4 | 16.9 (1.1) | 16.9 (1.3) | 17.0 (1.4)
  Week 8 | 17.6 (1.3) | 17.5 (1.2) | 17.6 (1.3)
  Week 12 | 17.8 (1.3) | 17.8 (1.1) | 17.7 (1.2)

ADVERSE EVENTS:
Arm/Group | Feihe New Formula | Feihe Formula | Breast Feeding
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No